CLINICAL TRIAL: NCT02857504
Title: One Lung Ventilation: Double-lumen Tube With vs Without Carinal Hook
Brief Title: One Lung Ventilation: Double Lumen Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Lea Andjelkovic, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 137/02/15
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Double Lumen Tube
Keywords: double lumen tube; hook

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- double lumen tube with a hook (Other): The tube with the hook (after passing the bronchial cuff trough the vocal cords) was rotated for 180 degrees to the left and removed the stylet and when the hook passed the vocal cords, the tube was rotated for 90 degrees back to the right and push it into the bronchus. Following formula was used for the right depth (height (cm)/10 + 12 (cm)) of the tube without the hook. The tube with hook was inserted into the bronchus so that hook was placed on the carina and stopped.
  Interventions: Device: double lumen tube with a hook
- double lumen tube without a hook (Other): Tube without the hook was inserted with the following technique: after the bronchial cuff was passed the vocal cords, the stylet was removed and the tube was rotated 90 st towards left.
  Interventions: Device: double lumen tube without a hook

INTERVENTIONS:
Device: double lumen tube with a hook — The tube with the hook (after passing the bronchial cuff trough the vocal cords) was rotated for 180 degrees to the left and removed the stylet and when the hook passed the vocal cords, the tube was rotated for 90 degrees back to the right and push it into the bronchus. Following formula was used for the right depth (height (cm)/10 + 12 (cm)) of the tube without the hook. The tube with hook was inserted into the bronchus so that hook was placed on the carina and stopped.
  Arms: double lumen tube with a hook
Device: double lumen tube without a hook — Tube without the hook was inserted with the following technique: after the bronchial cuff was passed the vocal cords, the stylet was removed and the tube was rotated 90 st towards left.
  Arms: double lumen tube without a hook

SUMMARY:
One lung ventilation (OLV) has become a standard procedure for the vast majority of interventions in pulmonary surgery. It is used in both techniques: thoracotomy and videothoracoscopy (VATS).

OLV can be provided by double lumen tube (DLT) with or without the hook. In our study the investigators want to find out if there is any advantage with one or another.

DETAILED DESCRIPTION:
One lung ventilation (OLV) has become a standard procedure for the vast majority of interventions in pulmonary surgery. It is used in both techniques: thoracotomy and videothoracoscopy (VATS)(1).

OLV can be provided by double lumen tube (DLT) or bronchial blocker. There are advantages and disadvantages of both techniques, but DLT is more recommended because it allows total emptying of the operated lung. Air and secretion can be aspirated through the wide lumen of the tube during the surgery (2, 3).

There are many kinds of DLT which differ according to shape and material. Most commonly used are left sided DLT which are placed into left main bronchus and right or left lungs can be closed or emptied. Left sided tube have a hook which is placed on the carina to prevent displacement of the tube. There are also DLT without the hook which are more gentle and easier to place in the left main bronchus (4,5). After the insertion of the left tube without the hook, bronchoscopy is recommended to check the position of the tube (6,7,8,9).

Some severe complications (injury of the bronchial tree) after insertion of the hooked tube are found in the literature (10). The investigators have published such complication from our experience (11).

Each anesthesiologist decides individually which kind of DLT to use as there are no studies which have objectivised the advantage of either technique. There is only one study where they have compared both techniques but they have found no difference. That is why the investigators decided to study which technique is better so this can be included in our standard operative procedure.

ELIGIBILITY:
Inclusion Criteria:

* planned thoracotomy or VATS surgical technique
* with ASA (American Society of Anesthesiologist) physical status 1-3.

Exclusion Criteria:

* ASA>3,
* severe heart illness (NYHA >3),
* severe pulmonary obstructive disease (FEV1<40%),
* neurologic disorders and
* patients with other respiratory or lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
intubation | intraoperative
  The time needed for tube insertion (time from seeing the vocal cords to final position of the tube) was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Result] Campos JH. Lung isolation techniques for patients with difficult airway. Curr Opin Anaesthesiol. 2010 Feb;23(1):12-7. doi: 10.1097/ACO.0b013e328331e8a7. PMID 19752725
- [Result] Pedoto A. How to choose the double-lumen tube size and side: the eternal debate. Anesthesiol Clin. 2012 Dec;30(4):671-81. doi: 10.1016/j.anclin.2012.08.001. PMID 23089502
- [Result] Hofmann HS, Rettig G, Radke J, Neef H, Silber RE. Iatrogenic ruptures of the tracheobronchial tree. Eur J Cardiothorac Surg. 2002 Apr;21(4):649-52. doi: 10.1016/s1010-7940(02)00037-4. PMID 11932162
- [Result] Prunet B, Lacroix G, Asencio Y, Cathelinaud O, Avaro JP, Goutorbe P. Iatrogenic post-intubation tracheal rupture treated conservatively without intubation: a case report. Cases J. 2008 Oct 22;1(1):259. doi: 10.1186/1757-1626-1-259. PMID 18945364
- [Result] Klein U, Karzai W, Bloos F, Wohlfarth M, Gottschall R, Fritz H, Gugel M, Seifert A. Role of fiberoptic bronchoscopy in conjunction with the use of double-lumen tubes for thoracic anesthesia: a prospective study. Anesthesiology. 1998 Feb;88(2):346-50. doi: 10.1097/00000542-199802000-00012. PMID 9477054
- [Result] Slinger PD. Fiberoptic bronchoscopic positioning of double-lumen tubes. J Cardiothorac Anesth. 1989 Aug;3(4):486-96. doi: 10.1016/s0888-6296(89)97987-8. PMID 2520925
- [Result] Cohen E. Double-lumen tube position should be confirmed by fiberoptic bronchoscopy. Curr Opin Anaesthesiol. 2004 Feb;17(1):1-6. doi: 10.1097/00001503-200402000-00002. PMID 17021522
- [Result] Fitzmaurice BG, Brodsky JB. Airway rupture from double-lumen tubes. J Cardiothorac Vasc Anesth. 1999 Jun;13(3):322-9. doi: 10.1016/s1053-0770(99)90273-2. No abstract available. PMID 10392687
- [Result] Dumans-Nizard V, Parquin JF, Moyer JD, Dreyfus JF, Fischler M, Le Guen M. Left double-lumen tube with or without a carinal hook: A randomised controlled trial. Eur J Anaesthesiol. 2015 Jun;32(6):418-24. doi: 10.1097/EJA.0000000000000201. PMID 25489763